CLINICAL TRIAL: NCT01469351
Title: Neurodegenerative Changes in Alzheimer's Disease: Identifying Potential Effects of Liraglutide on Degenerative Changes
Brief Title: Identifying Potential Effects of Liraglutide on Degenerative Changes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-000794-31
Record Dates: First submitted 2011-11-01; First posted 2011-11-10 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Alzheimers Disease
Keywords: Alzheimers disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug (Active Comparator): the GLP-1 receptor analog liraglutide is the active drug. The dose is 1.8mg daily
  Interventions: Drug: Liraglutide
- placebo (Placebo Comparator): non active intervention
  Interventions: Drug: non-active study drug

INTERVENTIONS:
Drug: Liraglutide — Liraglutide (Victoza ®), human GLP-1 analog produced using recombinant DNA technology in saccharomyces cerevisiae. Victoza ® is registered and approved for the treatment of type 2 diabetes.
  Victoza ® stimulates glucose-dependent insulin secretion from β-cells and inhibits glucagon secretion, slows ventricle emptying and reduces body weight and body fat mass by affecting appetite regulation.
  Form of administration: Liraglutide is a clear injection fluid, which comes in a prefilled disposable pen.
  1 ml contains 6 mg of liraglutide in sterile water. There is added disodium phosphate and propylene glycol and the preservative phenol. A filled pen contains 18mg liraglutide in 3ml. NovoFine® needles are used.
  Arms: Drug
Drug: non-active study drug — placebo
  Arms: placebo

SUMMARY:
Today Alzheimers disease can not be cured. Animal experiments have shown that the hormone GLP-1 can improve memory in Alzheimer-prone mice.

The investigators hypothesis is that a 6-month treatment with the GLP-1 receptor stimulating drug liraglutide will reduce the intracerebral amyloid deposition in the central nervous system (CNS) in patients with Alzheimer's disease (AD) and thereby reduce the clinical symptoms of the disease.

DETAILED DESCRIPTION:
The incidences of both type 2 diabetes (DM-2) and Alzheimer's disease (AD) have increased during the last years, resulting in an increase in morbidity and mortality. DM-2 is a risk factor for both AD and vascular dementia. In addition, an increased incidence of DM-2 in Alzheimer's patients has been observed. The understanding of the underlying mechanism behind this linkage is so far very sparse.

In both diseases premature cell degeneration develops. DM-2 is characterized by a loss of β-cell function and β cell mass in the pancreas, whereas AD shows a loss of neuronal function as well as neuronal cell death. General metabolic risk factors such as hyperglycemia and hypercholesterolemia are evident in both diseases.

Glucagon-like-peptide-1 (GLP-1) is an incretin hormone with numerous documented effects on the glycaemic response. It is released as a response to food ingestion and consequently exerts a glucose-dependent stimulation of insulin secretion while inhibiting glucagon secretion. In animal experiments as well as cell experiments β-cell neogenesis, growth and differentiation are stimulated by GLP-1, and inhibition of β-cell apoptosis has been demonstrated in cell studies. In addition to α- and β-cells of the pancreas, GLP-1 receptors (GLP-1R) have been localized to the CNS, where GLP-1R are distributed corresponding to the hypothalamus and hippocampus. Experimental investigations on mice where GLP-1 was given intra-cerebroventricularly, GLP-1R stimulation reduced nerve cell damage caused by neurotoxic stimuli. Furthermore, GLP-1R stimulation in hippocampus induced learning ability and memory and it has been shown that GLP-1R stimulation leeds to neurite outgrowth and protects against nerve cell apoptosis.

In connection with hyperinsulinaemia in early stages of DM-2, studies suggest that stimulation of insulin receptors represented in the brain produce an increased level of β-amyloid and an increased number of neurofibrillary tangles. AD is pathologically characterized by an increased level of β-amyloid as well as an increased number of neurofibrillar tangles. Accumulation of β-amyloid in the brain is localized to areas with cognitive functions. A recent animal experimental work has shown reduced memory in GLP-1 receptor KO mice and mentions the lack of a possible neuroprotective effect as a potential explanation for the observation. In studies of humans a worsening of the cognitive functions has been shown to be associated with dementia and DM-2, even though an actual causal relation has not yet been found. The investigators have recently shown that GLP-1 has a neuroprotective function in patients with DM-2.

Positron emission tomography (PET) scanning has been well evaluated in clinical demonstration of CNS changes following AD including changes in amyloid deposits.

Presently there are no registered drugs which change the deposition of amyloid and there are no drugs with convincing effect on the progression of the disease in patients with Alzheimer's. Moreover the drugs which have been marketed for treatment have a disadvantageous side effect profile. Besides insulin, β-cells secrete amylin, amyloid or IAPP (islet amyloid polypeptide) and these thus share certain characteristics with β-amyloid. Previously IAPP was considered to be non-toxic but recent studies have indicated a possible conversion to toxic β-amyloid.

The insulin-producing β-cells have been found to be characterized by accumulation of amyloid in several DM-2 models. A recent study with treatment with DPP-4 inhibitors (increasing endogenous GLP-1) improved glucose tolerance, increased GLP-1 levels and normalized the topography of the islets of Langerhans in a mouse model with β cell specific over expression of human amyloid.

The investigators hypothesis is that a 26 week treatment with the GLP-1 receptor stimulating pharmaceutical liraglutide will reduce the intracerebral amyloid deposition in the CNS in patients with Alzheimer's disease, as demonstrated by PET.

The investigators aim is that this clinical study will be able to give new information about the effect of the GLP-1 axis in the CNS and explore the potential for treatment of large groups of patients who cannot be offered effective drugs today. Altogether the results from the studies will contribute to the development of future treatment options for AD.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent before study-related activity
* Adult competent persons
* Diagnosed with diagnosed Alzheimer's disease. With a MMSE score between 18-21 the diagnosis should be entirely based on the clinic, while diagnosis by MMSE with a score > 22 should be diagnosed by spinal puncture
* Age ≥ 50 years and ≤ 80 years
* Caucasians

Exclusion Criteria:

* Diabetes mellitus
* Clinically significant liver (s-ALT > 2 times upper reference or creatinine-clearance < 30 mL / min, assessed on Cockcroft-Gault normogram)
* Clinically significant anemia
* Other clinically relevant abnormal biochemical value
* Current or former presence of one of the following diseases with clinical relevance:

  1. another CNS-illness other than diagnosed depression treated with SSRI or SSRI similar drugs.
  2. liver disease
  3. kidney disease
  4. endocrinological disease other than well controlled hypothyroidism
* Current or history of chronic or acute pancreatitis
* Any disease which the investigators believe may affect the study
* Patients treated with TCA or neuroleptics
* Known abuse of alcohol or drugs
* Known allergy to liraglutide or any of the other components (disodium phosphate dihydrate, propylene glycol and phenol)
* Participation in a clinical trial less than 3 months before inclusion in this study
* Persons who within a period of the last 2 years have participated in scientific experiments involving the use of isotopes, or who have had greater diagnostic tests performed using applied ionizing radiation
* If patients are treated with SSRI or SSRI similar drugs or antihypertensives this treatment should be stable
* Claustrophobia or other missing cooperation
* Severe overweight > 130kg
* Ferro-magnetic prosthesis, pacemaker or other metals incorporated in the body
* Significant abnormities in the brain detected by MR scanning

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
PIB PET scan | PIB PET-scan at baseline and after 26 weeks
  Primarily to investigate whether 26 weeks of treatment with GLP-1 receptor liraglutide (Victoza ®) will change the intra-cerebral amyloid deposit in the CNS in patients with Alzheimer's disease assessed by PIB PET scan.

SECONDARY OUTCOMES:
Neuro-psychological tests | At baseline, after 12 weeks and after 26 weeks
  To validate the cognitive functions using specific neuro-psychological test battery before and after treatment with liraglutide/placebo.
FDG PET Scan | FDG PET-scan at baseline and after 26 weeks
  To examine changes in glucose uptake in the CNS by FDG PET scan before and after 6 months of treatment with liraglutide/placebo

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte Brock, MD phD, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Aarhus, Denmark

REFERENCES:
- [Background] Abbas T, Faivre E, Holscher C. Impairment of synaptic plasticity and memory formation in GLP-1 receptor KO mice: Interaction between type 2 diabetes and Alzheimer's disease. Behav Brain Res. 2009 Dec 14;205(1):265-71. doi: 10.1016/j.bbr.2009.06.035. Epub 2009 Jun 30. PMID 19573562
- [Background] Cole AR, Astell A, Green C, Sutherland C. Molecular connexions between dementia and diabetes. Neurosci Biobehav Rev. 2007;31(7):1046-63. doi: 10.1016/j.neubiorev.2007.04.004. Epub 2007 Apr 24. PMID 17544131
- [Background] Dimou E, Booij J, Rodrigues M, Prosch H, Attems J, Knoll P, Zajicek B, Dudczak R, Mostbeck G, Kuntner C, Langer O, Bruecke T, Mirzaei S. Amyloid PET and MRI in Alzheimer's disease and mild cognitive impairment. Curr Alzheimer Res. 2009 Jun;6(3):312-9. doi: 10.2174/156720509788486563. PMID 19519314
- [Background] During MJ, Cao L, Zuzga DS, Francis JS, Fitzsimons HL, Jiao X, Bland RJ, Klugmann M, Banks WA, Drucker DJ, Haile CN. Glucagon-like peptide-1 receptor is involved in learning and neuroprotection. Nat Med. 2003 Sep;9(9):1173-9. doi: 10.1038/nm919. Epub 2003 Aug 17. PMID 12925848
- [Derived] Muscogiuri G, DeFronzo RA, Gastaldelli A, Holst JJ. Glucagon-like Peptide-1 and the Central/Peripheral Nervous System: Crosstalk in Diabetes. Trends Endocrinol Metab. 2017 Feb;28(2):88-103. doi: 10.1016/j.tem.2016.10.001. Epub 2016 Oct 27. PMID 27871675
- [Derived] Gejl M, Gjedde A, Egefjord L, Moller A, Hansen SB, Vang K, Rodell A, Braendgaard H, Gottrup H, Schacht A, Moller N, Brock B, Rungby J. In Alzheimer's Disease, 6-Month Treatment with GLP-1 Analog Prevents Decline of Brain Glucose Metabolism: Randomized, Placebo-Controlled, Double-Blind Clinical Trial. Front Aging Neurosci. 2016 May 24;8:108. doi: 10.3389/fnagi.2016.00108. eCollection 2016. PMID 27252647
- [Derived] Egefjord L, Gejl M, Moller A, Braendgaard H, Gottrup H, Antropova O, Moller N, Poulsen HE, Gjedde A, Brock B, Rungby J. Effects of liraglutide on neurodegeneration, blood flow and cognition in Alzheimer s disease - protocol for a controlled, randomized double-blinded trial. Dan Med J. 2012 Oct;59(10):A4519. PMID 23158895
- See also: information about Alzheimers disease — http://alzheimers.org